CLINICAL TRIAL: NCT02686580
Title: Feasibility Study to Assess the Early Use of Porcine Cross-linked Collagen Paste in Cryptoglandular Anorectal Fistulas
Acronym: FIX-IT1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit participants for this study
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1510144
Record Dates: First submitted 2015-12-01; First posted 2016-02-19 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2016-02

CONDITIONS: Anorectal Abscess; Fistula in Ano
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collagen paste (Experimental): Injection of Permacol Collagen paste into the fistula tract.
  Interventions: Biological: Collagen paste

INTERVENTIONS:
Biological: Collagen paste — Permacol cross-linked collagen paste, 2.5-3.5 mls to be injected into the MRI defined fistula tracts 7-10 days following drainage of the anorectal abscess.

SUMMARY:
This study is designed to assess the effectiveness of porcine cross-linked collagen paste for the treatment of patients with ano-rectal abscess with underlying cryptoglandular fistula in ano.

DETAILED DESCRIPTION:
Most anal fistulae are thought to arise as a result of the infection of anal glands. This infection frequently presents as an anorectal abscess which requires drainage of the abscess under a general anaesthetic. Abscess and fistula should be considered as the acute and chronic phase of the same anorectal infection.The abscess represents the acute inflammatory event, whereas the fistula is representative of the chronic process. At the time of drainage of the anorectal abscess, the underlying fistulas frequently go undetected. As a result, patients present with a fistula in ano several months later.

In this study, the investigators aim to identify the underlying fistula in patients with a perianal abscess with the help of an MRI Scan done in the acute setting. Participants with a confirmed fistula on the MRI scan have their abscess treated as per convention. However, a repeat examination under anaesthetic is performed 7-'10 days later when the fistula tract is identified and treated with injection of the porcine collagen paste into the fistula tract. Participants are followed up clinically and radiologically to assess the effectiveness of the intervention.

ELIGIBILITY:
* Inclusion Criteria:

  o Clinical diagnosis of Cryptoglandular fistula in ano.
* Exclusion Criteria:

  * Insulin dependent diabetes
  * Thyroid disease
  * Fistula secondary to Crohn's disease/Ulcerative Colitis
  * Clinical or radiological evidence of secondary tracts.
  * Complex fistula tracts on MRI scan such as Horseshoe fistula, anorectal-vaginal fistula
  * Patients refusing informed consent for admission to the study.
  * Previous fistulotomy/fistulectomy
  * Pregnancy
  * Patients unable to consent
  * Patients not suitable for MRI scan those with- Cochlear implant, Permanent pacemaker, Implanted metal work, Aneurysm clips, Claustrophobia, Metallic foreign body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Fistula Healing rate at 3 months | 3 months
  Healing of fistula as evidenced by MRI of the ano-rectum.
Fistula Healing Rate at 12 months | 12 months
  This will be assessed by a telephonic questionnaire at 12 months following intervention

SECONDARY OUTCOMES:
Complication rate | 12 months
  Any complications resulting from participation in the the trial will be assessed on clinical and telephonic follow up. Clavien and Dindo Classification will be used to assess the severity of complications.
Faecal Incontinence questionnaire (Wexner) | At recruitment, 7-10 days, 6 weeks and 6 months
  To assess any adverse impact of intervention on continence
Faecal Incontinence quality of life questionnaire (FIQL) | At recruitment, 7-10 days, 6 weeks and 6 months
  To assess the impact on the quality of life of the participants
Pain Score | At recruitment, 7-10 days, 6 weeks and 6 months
  Visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Neil J Smart, MBBS PhD FRCS, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Undecided